CLINICAL TRIAL: NCT00886808
Title: A Phase I, Open-Label, Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of iCo-007 Intravitreal Injection in Subjects With Diffuse Diabetic Macular Edema
Brief Title: Safety Study of iCo-007 Intravitreal Injection to Treat Diabetic Macular Edema
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: iCo Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-007-01-DME
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Diffuse Diabetic Macular Edema
Keywords: DME, Diabetic Retinopathy, Diabetic Macular Edema
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): 110 microgram dose of iCo-007 Intravitreal Injection
  Interventions: Drug: iCo-007 Intravitreal Injection
- 2 (Experimental): 350microgram dose of iCo-007 Intravitreal Injection
  Interventions: Drug: iCo-007 Intravitreal Injection
- 3 (Experimental): 700microgram dose of iCo-007 Intravitreal Injection
  Interventions: Drug: iCo-007 Intravitreal Injection
- 4 (Experimental): 1,000microgram dose of iCo-007 Intravitreal Injection
  Interventions: Drug: iCo-007 Intravitreal Injection

INTERVENTIONS:
Drug: iCo-007 Intravitreal Injection — single dose iCo-007 Intravitreal Injection

SUMMARY:
The goal of the study is to evaluate the safety and tolerability of 4 different doses of iCo-007 Intravitreal Injection in patients with diffuse diabetic macular edema.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women 18 years of age or older
2. Confirmed diagnosis of diabetes mellitus type I or II (both, insulin or non-insulin dependent)
3. Subjects who have moderate to severe non-proliferative diabetic retinopathy (NPDR), as defined by ETDRS criteria, and diffuse DME within 300 microns from the center of the macula in the study eye (with or without cystoid changes) confirmed by FA.
4. Retinal thickness must be at least 250 microns in the central subfield, as shown by OCT
5. Best-corrected visual acuity between 60 and 15 letters measured with ETDRS charts (approximately 20/63 to 20/500 with Snellen charts)
6. Woman of child-bearing potential must not be pregnant or lactating, must have a negative pregnancy test at screening (serum). Both men and women are required to practice an adequate method of birth control
7. Able and willing to sign an approved informed consent form and return for all scheduled study visits

Exclusion Criteria:

1. Subjects with macular or perimacular edema secondary to an etiology other than diabetes mellitus
2. Subjects with concurrent retinal diseases or conditions in the study eye (including conditions requiring urgent PRP), glaucoma (or ocular hypertension), retinal vascular occlusion, exudative age-related macular degeneration (drusen permitted), tear (rip) of the retinal pigment epithelium, a vitelliform-like lesion of the outer retina (e.g. pattern dystrophies or basal laminar drusen), idiopathic parafoveal telangiectasis or retinal-lesion anastomosis
3. Subjects who have any additional ocular disease or condition which could compromise treatment safety, visual acuity or interfere with assessment of the macular edema, such as ocular inflammation, amblyopia, anterior ischemic optic neuropathy, media opacity, cataract
4. Subjects who have diffuse DME with severe capillary non-perfusion (avascular zone diameter >1,000 microns)
5. Allergy to fluorescein dye
6. Subjects who had intraocular surgery, photocoagulation, intravitreal or subfoveal injection, topical or systemic steroids or who received any experimental treatment as part of another clinical trial within the last 3 months of the study start (in case of Anecortave within the last 6 months, any panretinal photocoagulation prior to study start)
7. Subjects with uncontrolled diabetes (glycosylated hemoglobin Hb A1c >12%)
8. Subjects with systolic blood pressure higher than 180 mm Hg or diastolic above 100 mm Hg, with or without anti-hypertensive treatment
9. Subjects with congestive heart disease or any unstable cardiac condition
10. Subjects with clinically significantly impaired renal function (serum creatinine >2.0 mg/dL) and/or moderate to severe hepatic impairment (subjects with >2.5 times the upper limit of the normal range for aspartate transaminase [AST], alanine transaminase [ALT], or total bilirubin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-02; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of 4 dose levels of intravitreal administration of iCo-007. | At multiple points after injection up to and including 6 months

SECONDARY OUTCOMES:
To assess the systemic pharmacokinetics of iCo-007 after intravitreal administration. To assess change in retinal thickness relative to baseline as determined by OCT. To assess change in best corrected visual acuity relative to baseline. | At multiple points after injection up to and including 6 months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Retina-Vitreous Associates Medical Group, Los Angeles, California
  - Bascom Palmer Eye Institute, Miami, Florida
  - Duke Eye Center, Durham, North Carolina
  - Valley Retina Institute, McAllen, Texas